CLINICAL TRIAL: NCT03627091
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled, Parallel-group Efficacy and Safety Study of SHP647 as Maintenance Therapy in Subjects With Moderate to Severe Crohn's Disease (CARMEN CD 307)
Brief Title: Efficacy and Safety Study of Ontamalimab as Maintenance Treatment in Participants With Moderate to Severe Crohn's Disease (CARMEN CD 307)
Acronym: CARMEN CD 307
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision to discontinue the SHP647 (ontamalimab) clinical trial development program for inflammatory bowel diseases (IBD) early.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHP647-307; 2017-000617-23 (EudraCT Number)
Record Dates: First submitted 2018-07-24; First posted 2018-08-13 (Actual); Results first posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease
MeSH Terms: conditions — Crohn Disease | interventions — ontamalimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ontamalimab 25 mg (Experimental): Participants will receive 25 mg of ontamalimab subcutaneous (SC) injection using a prefilled syringe once every 4 weeks for 52 weeks; starting at Day/Week 1 Baseline Visit (Week 16 of the SHP647-305 [NCT03559517] or SHP647-306 [NCT03566823]).
  Interventions: Drug: Ontamalimab
- Ontamalimab 75 mg (Experimental): Participants will receive 75 mg of ontamalimab SC injection using a prefilled syringe once every 4 weeks for 52 weeks; starting at Day/Week 1 Baseline Visit (Week 16 of the SHP647-305 [NCT03559517] or SHP647-306 [NCT03566823]).
  Interventions: Drug: Ontamalimab
- Placebo (Placebo Comparator): Participants will receive placebo matched with ontamalimab SC injection using prefilled syringe once every 4 weeks for 52 weeks; starting at Day/Week 1 Baseline Visit (Week 16 of the SHP647-305 [NCT03559517] or SHP647-306 [NCT03566823]).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ontamalimab — SC injection of 25 mg or 75 mg ontamalimab will be administered using a prefilled syringe.
  Other Names: SHP647; PF-00547659
  Arms: Ontamalimab 25 mg; Ontamalimab 75 mg
Other: Placebo — SC injection of placebo matched with ontamalimab will be administered using a prefilled syringe.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ontamalimab as maintenance treatment in participants with moderate to severe Crohn's disease (CD).

ELIGIBILITY:
Inclusion Criteria:

* Participants and/or their parent or legally authorized representative (LAR) must have an understanding, ability, and willingness to fully comply with study procedures and restrictions.
* Participants must be able to voluntarily provide written, signed, and dated (personally or via a LAR) informed consent and/or assent, as applicable, to participate in the study.
* Participants must have completed the 16-week induction treatment period from study SHP647-305 (NCT03559517) or SHP647-306 (NCT03566823) and met the following criteria at baseline in maintenance study SHP647-307:

  1. Meet endoscopic response criteria of a reduction in SES-CD from induction studies SHP647-305 (NCT03559517) or SHP647-306 (NCT03566823) baseline by greater than or equal to >=25% at Week 16 of induction studies SHP647-305 (NCT03559517) or SHP647-306 (NCT03566823) or
  2. Meet at least 1 of the following 4 criteria at baseline in maintenance study SHP647-307, in addition to no worsening of endoscopic score as measured by SES-CD relative to induction studies SHP647-305 (NCT03559517) or SHP647-306 (NCT03566823) baseline:
* Achieving clinical remission as determined by meeting the criteria for clinical remission using the 2-item PRO, that is, 2-item PRO sub scores of average worst daily abdominal pain <=3 (based on 11-point NRS) over the 7 most recent days* and average daily stool type frequency <=2 of type 6/7 (very soft stools/liquid stools) as shown in the Bristol Stool Form Scale (BSFS) over the 7 most recent days*.
* A decrease of at least 100 points in CDAI score (CDAI-100) from induction studies baseline.
* A decrease of >=30% and at least 2 points from induction studies baseline in the average daily worst abdominal pain over the 7 most recent days*, with the average daily stool frequency of type 6/7 (very soft stools/liquid stools) either: (i) not worsening from induction studies baseline and/or (ii) meeting the criteria for clinical remission, that is, 2-item PRO subscore of average daily stool frequency <=2 of type 6/7 (very soft stools/liquid stools) as shown in the BSFS over the 7 most recent days*.
* A decrease of >=30% from induction studies SHP647-305 (NCT03559517) or SHP647-306 (NCT03566823) baseline in the average daily stool frequency of type 6/7 (very soft stools/liquid stools) as shown in the BSFS over the 7 most recent days*, with the average daily worst abdominal pain either: (i) not worsening from induction studies SHP647-305 (NCT03559517) or SHP647-306 (NCT03566823) baseline and/or (ii) meeting the criteria for clinical remission, that is, 2-item PRO sub score of average worst daily abdominal pain <=3 (based on 11-point NRS) over the 7 most recent days*.

  *Note: The 7 days may or may not be contiguous during the 10 days of data collection before colonoscopy preparation, depending on days to be excluded because of missing data. If fewer than 7 days are available, the criterion will be calculated on all available most recent 6 or 5 days. If fewer than 5 days are available, the criterion will be treated as missing.
* Participants receiving any treatments for CD are eligible provided they have been, and are anticipated to be, on a stable dose for the designated period of time.

Exclusion Criteria:

* Participants who had major protocol deviations (as determined by the sponsor) in induction studies SHP647-305 (NCT03559517) or SHP647-306 (NCT03566823).
* Participants who permanently discontinued investigational product because of an AE, regardless of relatedness to investigational product, in induction studies SHP647-305 (NCT03559517) or SHP647-306 (NCT03566823).
* Participants who are likely to require surgery for CD during the study period, except minor interventions (eg, seton placement for anal fistulas).
* Participants are females who became pregnant during induction studies SHP647-305 (NCT03559517) or SHP647-306 (NCT03566823), females who are lactating, females who are planning to become pregnant during the study period, or males or females of childbearing potential not agreeing to continue acceptable contraception methods (ie, highly effective methods for female participants and medically appropriate methods for male participants) through the conclusion of study participation.
* Participants who do not agree to postpone donation of any organ or tissue, including male participants who are planning to bank or donate sperm and female participants who are planning to harvest or donate eggs, for the duration of the study and through 16 weeks after last dose of investigational product.
* Participants who, in the opinion of the investigator or the sponsor, will be uncooperative or unable to comply with study procedures.
* Participants who have developed obstructive colonic stricture, or enterovesical or enterovaginal fistulae during the induction study SHP647-305 (NCT03559517) or SHP647-306 (NCT03566823).
* Participants who have a newly diagnosed malignancy or recurrence of malignancy (other than resected cutaneous basal cell carcinoma, squamous cell carcinoma, or carcinoma in situ of the uterine cervix that has been treated with no evidence of recurrence).
* Participants who have developed any major illness/condition or evidence of an unstable clinical condition (example [eg,] renal, hepatic, hematologic, gastrointestinal (except disease under study), endocrine, cardiovascular, pulmonary, immunologic [eg, Felty's syndrome], or local active infection/infectious illness) that, in the investigator's judgment, will substantially increase the risk to the participant if he or she participates in the study.
* Participants with any other severe acute or chronic medical or psychiatric condition or laboratory or ECG abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Participants with known exposure to Mycobacterium tuberculosis (TB) since testing at screening in induction studies SHP647-305 (NCT03559517) or SHP647-306 (NCT03566823) and who have been advised to require treatment for latent or active disease but who are without a generally accepted course of treatment.
* Participants with any of the following abnormalities in hematology and/or serum chemistry profiles during the evaluation of the last visit in the induction studies SHP647-305 (NCT03559517) or SHP647-306 (NCT03566823). If the results are considered by the investigator to be transient and inconsistent with the participant's clinical condition, may be repeated once prior to enrollment in Study SHP647-307.

  1. Alanine aminotransferase (ALT) and aspartate aminotransferase levels >= 3.0 × the upper limit of normal (ULN).
  2. Total bilirubin level >=1.5 × ULN or >2.0 × ULN if the participant has a known documented history of Gilbert's syndrome.
  3. Hemoglobin level <=80 gram per liter (g/L) (8.0 gram per deciliter [g/dL]).
  4. Platelet count <=100 × 10^9/L (100,000 cells per cubic millimeter [mm^3]) or >=1000 × 10^9/L (1,000,000 cells/mm^3).
  5. White blood cell count <=3.5 × 10^9/L (3500 cells/mm^3).
  6. Absolute neutrophil count<2 × 10^9/L (<2000 cells/mm^3)
  7. Serum creatinine level >1.5 × ULN or estimated glomerular filtration rate <30 milliliter per minute (mL/min)/1.73 m^2 based on the abbreviated Modification of Diet in Renal Disease Study Equation.

     * Note: If platelet count is <150,000 cells/mm^3, a further evaluation should be performed to rule out cirrhosis, unless another etiology has already been identified.
* Participants who are investigational site staff members or relatives of those site staff members or participants who are sponsor employees directly involved in the conduct of the study.
* Participants who are participating in other investigational studies (other than induction studies SHP647-305 [NCT03559517] or SHP647-306 [NCT03566823]) or plan to participate in other investigational studies during this study.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (280):
- United States (72):
  - Arizona Digestive Health Mesa - East, Mesa, Arizona
  - Elite Clinical Studies - Phoenix - Clinedge - PPDS, Phoenix, Arizona
  - CATS Research Center - University of Arizona, Tucson, Arizona
  - Atria Clinical Research - Clinedge - PPDS, Little Rock, Arkansas
  - Advanced Research Center, Anaheim, California
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - OM Research LLC - Lancaster - ClinEdge - PPDS, Lancaster, California
  - Alliance Clinical Research-(Vestavia Hills), Poway, California
  - Inland Empire Liver Foundation, Rialto, California
  - Care Access Research, San Pablo, San Pablo, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Asthma and Allergy Associates PC - CRN - PPDS, Colorado Springs, Colorado
  - Renaissance Research Medical Group, INC, Cape Coral, Florida
  - Gastro Florida, Clearwater, Florida
  - Advanced Clinical Research Network, Coral Gables, Florida
  - Alliance Medical Research LLC, Coral Springs, Florida
  - SIH Research, Kissimmee, Florida
  - Hi Tech and Global Research, LLc, Miami, Florida
  - Sanchez Clinical Research, Inc, Miami, Florida
  - Crystal Biomedical Research, Miami Lakes, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Pharma Research International Inc, Naples, Florida
  - Omega Research Consultants LLC - Clinedge - PPDS, Orlando, Florida
  - Accel Research Sites - St. Petersburg - ERN - PPDS, Pinellas Park, Florida
  - East Coast Institute for Research, LLC, Saint Augustine, Florida
  - DBC Research, Tamarac, Florida
  - Bayside Clinical Research - New Port Richey, Tampa, Florida
  - Atlanta Gastroenterology Specialists, PC, Atlanta, Georgia
  - Infinite Clinical Trials, Atlanta, Georgia
  - Atlanta Center For Gastroenterology PC, Decatur, Georgia
  - Loretto Hospital, Chicago, Illinois
  - IL Gastroenterology Group, Gurnee, Illinois
  - Laporte County Institute For Clinical Research, Michigan City, Indiana
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Gastroenterology Associates of Hazard, Hazard, Kentucky
  - CroNOLA, LLC., Houma, Louisiana
  - Clinical Trials of SWLA, LLC, Lake Charles, Louisiana
  - DelRicht Clinical Research, LLC - ClinEdge - PPDS, New Orleans, Louisiana
  - Louisiana Research Center LLC, Shreveport, Louisiana
  - Commonwealth Clinical Studies LLC, Brockton, Massachusetts
  - Winchester Gastroenterology Associates, Winchester, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, Chesterfield, Michigan
  - National Clinical, LLC, Hamtramck, Michigan
  - Gastroenterology Associates of Western Michigan, PLC, Wyoming, Michigan
  - Mayo Clinic Health System - PPDS, Duluth, Minnesota
  - Minnesota Gastroenterology PA, Saint Paul, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Encompass Care, North Las Vegas, Nevada
  - New York Total Medical Care PC, Brooklyn, New York
  - NYU Langone Long Island Clinical Research Associates, Great Neck, New York
  - Southtowns Gastroenterology, PLLC, Orchard Park, New York
  - Piedmont Healthcare, Statesville, North Carolina
  - Consultants For Clinical Research Inc, Cincinnati, Ohio
  - Consultants For Clinical Research Inc, Fairfield, Ohio
  - Penn State Hershey Medical Group, State College, Pennsylvania
  - Digestive Disease Associates, Wyomissing, Pennsylvania
  - Gastro One, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Advanced Gastroenterology-Union City, Union City, Tennessee
  - Northside Gastroenterology, Cypress, Texas
  - Digestive Health Associates of Texas, P.A.dba DHAT Research Institute, Garland, Texas
  - Precision Research Institute, LLC, Houston, Texas
  - Biopharma Informatic Inc., Houston, Texas
  - Southwest Clinical Trials, Houston, Texas
  - BI Research Center, Houston, Texas
  - Southern Star Research Institute LLC, San Antonio, Texas
  - Inquest Clinical Research/Coastal Gastroenterology Associates, PA - TDDC - PPDS, Webster, Texas
  - HP Clinical Research, Bountiful, Utah
  - Mid Atlantic Health Specialists, Galax, Virginia
- Argentina (2):
  - Fundación Favaloro, Buenos Aires
  - Hospital Privado Centro Médico de Córdoba, Córdoba
- Australia (6):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Mater Hospital Brisbane, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - St Vincents Hospital Melbourne - PPDS, Fitzroy, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Austria (4):
  - LKH-Universitätsklinikum Klinikum Graz, Graz, Styria
  - Klinikum Wels-Grieskirchen GmbH, Vienna, Vienna
  - Salzburger Landeskliniken, Salzburg
  - Medizinische Universitat Wien (Medical University of Vienna), Vienna
- Belgium (4):
  - Academisch Medisch Centrum Amsterdam, Bonheiden, Antwerpen
  - UZ Gent, Ghent, Oost-Vlaanderen
  - AZ Groeninge, Kortrijk, West-Vlaanderen
  - CHU Mouscron, Mouscron
- Clinical Center Banja Luka, Banja Luka, Bosnia and Herzegovina
- Bulgaria (9):
  - Acibadem City Clinic University Multiprofile Hospital for Active Treatment EOOD, Sofia, Sofia-Grad
  - Multiprofile Hospital for Active Treatment Eurohospital, Plovdiv
  - Second Multiprofile Hospital for Active Treatment Sofia, Sofia
  - Diagnostic and Consulting Center Aleksandrovska EOOD, Sofia
  - University Multiprofile Hospital for Active Treatment Sv Ivan Rilski EAD, Sofia
  - University Multiprofile Hospital for Active Treatment Tsaritsa Yoanna - ISUL EAD, Sofia
  - Medical Center Excelsior OOD - PPDS, Sofia
  - Medical Center Convex EOOD, Sofia
  - Diagnostic Consultative Centre Mladost - M OOD, Varna
- Colombia (2):
  - Fundación Valle Del Lili, Cali, Valle del Cauca Department
  - IPS Centro Médico Julián Coronel S.A.S. - PPDS, Cali
- Croatia (4):
  - University Hospital Center Zagreb, Zagreb, City of Zagreb
  - Opca bolnica Bjelovar, Bjelovar
  - Clinical Hospital Centre Osijek, Osijek
  - General Hospital Virovitica, Virovitica
- Estonia (2):
  - OÜ LV Venter, Pärnu
  - West Tallinn Central Hospital, Tallinn
- Germany (10):
  - Klinikum rechts der Isa der Technischen Universitaet Muenchen, Munich, Bavaria
  - Universitätsklinikum der RWTH Aachen, Aachen, North Rhine-Westphalia
  - Uniklinik Köln, Cologne, North Rhine-Westphalia
  - Gastro Campus Research GbR, Münster, North Rhine-Westphalia
  - Universitatsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
  - Universitatsklinikum Jena, Jena, Thuringia
  - Charité - Universitätsmedizin Berlin, Berlin
  - Gastroenterologische Facharztpraxis am Mexikoplatz, Berlin-Zehlendorf
  - Sana Klinikum Biberach, Biberach an der Riss
  - Universitätsklinikum Frankfurt, Frankfurt
- Greece (5):
  - Ippokrateio General Hospital of Athens, Athens, Attica
  - University General Hospital of Heraklion, Heraklion
  - Iatriko Palaiou Falirou, Paliao Faliro
  - University General Hospital of Patras, Pátrai
  - Euromedica - PPDS, Thessaloniki
- Hungary (8):
  - Bekes Megyei Kozponti Korhaz, Békéscsaba
  - Magyar Honvédség Egészségügyi Központ, Budapest
  - Pannónia Magánorvosi Centrum Kft, Budapest
  - ENDOMEDIX Kft., Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Mohacsi Korhaz, Mohács
  - Tolna Megyei Balassa János Kórház, Szekszárd
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- St Vincent's University Hospital, Dublin, Ireland
- Israel (4):
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center - PPDS, Jerusalem
  - Galilee Medical Center, Nahariya
  - Baruch Padeh Poriya Medical Center, Tiberias
- Italy (11):
  - Azienda Ospedaliera Mater Domini Di Catanzaro, Catanzaro, Calabria
  - Azienda Ospedaliero Universitaria Di Modena Policlinico, Modena, Emilia-Romagna
  - Fondazione Policlinico Universitario A Gemelli, Rome, Lazio
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - IRCCS Ospedale Sacro Cuore Don Calabria, Negrar, Veneto
  - A.O.U. Maggiore della Carità, Novara
  - Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia
  - La Sapienza-Università di Roma-Policlinico Umberto I, Roma
  - Istituto Clinico Humanitas, Rozzano (MI)
  - Ospedale Casa Sollievo Della Sofferenza IRCCS, San Giovanni Rotondo
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
- Japan (21):
  - Sapporo Medical University Hospital, Sapporo, Hokkaidô
  - Medical Corporation Aoyama Clinic, Kobe, Hyôgo
  - Hyogo College of Medicine, Nishinomiya-shi, Hyôgo
  - Jikei University Hospital, Minato-ku, Tokyo
  - Ome Municipal General Hospital, Ōme, Tokyo
  - Kunimoto Hospital, Asahikawa
  - Hidaka Coloproctology Clinic, Kurume-shi
  - Aichi Medical University Hospital, Nagakute
  - Nishinomiya Municipal Central Hospital, Nishinomiya
  - Onomichi General Hospital, Onomichi
  - Chiinkai Dojima General & Gastroenterology Clinic, Osaka
  - Kinshukai Infusion Clinic, Osaka
  - Yodogawa Christian Hospital, Osaka
  - Shiga University of Medical Science Hospital, Ōtsu
  - Toho University Sakura Medical Center, Sakura
  - Sapporo Higashi Tokushukai Hospital, Sapporo
  - Sapporo Tokushukai Hospital, Sapporo
  - Dokkyo Medical University Hospital, Shimotsuga-gun
  - Nihonbashi Egawa Clinic, Tokyo
  - Colo-Proctology Center Matsushima Clinic, Yokohama
  - Ishida Clinic of IBD and Gastroenterology, Ōita, Ôita
- Lebanon (2):
  - Al Zahraa University Hospital, Beirut
  - Hammoud Hospital University Medical Center, Saida
- Lithuania (2):
  - Vilnius University Hospital Santaros Klinikos, Vilnius
  - Vilnius City Clinical Hospital, Vilnius
- Mexico (7):
  - Investigacion Biomedica para el Desarrollo de Farmacos S.A. de C.V., Zapopan, Jalisco
  - Clinica de Higado y Gastroenterologia Integral, S.C., Cuernavaca, Morelos
  - JM Research S.C, Cuernavaca, Morelos
  - Accelerium, S. de R.L. de C.V., Monterrey, Nuevo León
  - Unidad de Atencion Medica e Investigacion en Salud, Mérida, Yucatán
  - Centro de Investigacion Clinica Acelerada, S.C., Distrito Federal
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
- Netherlands (2):
  - ETZ-Elisabeth, Tilburg, North Brabant
  - NWZ, location Alkmaar, Den Helder, North Holland
- New Zealand (3):
  - Dunedin Hospital, Dunedin, South Island
  - Wellington Hospital, Newtown, Wellington Region
  - Waikato Hospital, Hamilton
- Poland (29):
  - Vitamed Galaj i Cichomski sp.j., Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Gastromed Kopon Zmudzinski i Wspolnicy Sp.j.Specjalistyczne Centrum Gastrologii i Endoskopii Specj, Torun, Kuyavian-Pomeranian Voivodeship
  - Centrum Diagnostyczno - Lecznicze Barska sp. z o.o., Włocławek, Kuyavian-Pomeranian Voivodeship
  - Melita Medical, Wroclaw, Lower Silesian Voivodeship
  - Lexmedica, Wroclaw, Lower Silesian Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej CENTRUM MEDYCZNE Szpital Swietej Rodziny, Lódz, Lódzkie
  - Centrum Opieki Zdrowotnej Orkan-Med Stec-Michalska Sp. J., Lódz, Lódzkie
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Warsaw, Masovian Voivodeship
  - Niepubliczny Zakład Opieki Zdrowotnej VIVAMED, Warsaw, Masovian Voivodeship
  - Miedzyleski Szpital Specjalistyczny w Warszawie, Warsaw, Masovian Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok, Podlaskie Voivodeship
  - Endoskopia Sp. z o.o., Sopot, Pomeranian Voivodeship
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin, West Pomeranian Voivodeship
  - Szpital Uniwersytecki Nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Centrum Medyczne Czestochowa - PRATIA - PPDS, Częstochowa
  - Centrum Medyczne Gdynia - PRATIA - PPDS, Gdynia
  - NZOZ All Medicus, Katowice
  - Med Gastr Sp.z.o.o Sp.k, Lodz
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Twoja Przychodnia - Centrum Medyczne Nowa Sol, Nowa Sól
  - Clinical Research Center Spółka z Ograniczoną Odpowiedzialnością, Medic-R Spółka Komandytowa, Poznan
  - Centrum Medyczne Warszawa - PRATIA - PPDS, Rzeszów
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów
  - Sonomed Sp. z o.o., Szczecin
  - Centrum Zdrowia M D M, Warsaw
  - Centralny Szpital Kliniczny MSW, Warsaw
  - BioVirtus Centrum Medyczne, Warsaw
  - Samodzielny Publiczny Szpital Wojewodzki im. Papieza Jana Pawla II, Zamość
  - Szpital Specjalistyczny sw Lukasza - Oddzial Gastroenterologii, Gmina Końskie, Świętokrzyskie Voivodeship
- Portugal (3):
  - Hospital Senhora da Oliveira - Guimaraes, E.P.E, Guimarães
  - Hospital da Luz, Lisbon
  - Centro Hospitalar do Algarve - Hospital de Portimao, Portimão
- Romania (12):
  - Sana Monitoring SRL, Bucharest, București
  - Cluj-Napoca Emergency Clinical County Hospital, Cluj-Napoca, Cluj
  - Dr.Carol Davila Emergency University Central Military Hospital, Bucharest
  - Colentina Clinical Hospital, Bucharest
  - Prof. Dr. Matei Bals Institute of Infectious Diseases, Bucharest
  - Fundeni Clinical Institute, Bucharest
  - Centrul Medical Hifu Terramed Conformal S.R.L., Bucharest
  - Emergency University Hospital, Bucharest
  - Affidea Romania SRL, Constanța
  - Gastromedica SRL, Iași
  - Dr. Tirnaveanu Amelita Private Practice, Oradea
  - Dr. Goldis Gastroenterology Center SRL, Timișoara
- Russia (6):
  - Rostov State Medical University, Rostov-on-Don
  - St. Elizabeth Municipal Clinical Hospital, Saint Petersburg
  - Russian Medical Military Academy n.a. S.M. Kirov, Saint Petersburg
  - Medical University Reaviz, Samara
  - Private Healthcare Institution Clinical Hospital RZD-Medicina of Samara city, Samara
  - SHI Regional Clinical Hospital, Saratov
- Serbia (5):
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - University Clinical Center Nis, Niš
  - General Hospital Vrsac, Vršac
  - Clinical Hospital Center Zemun, Zemun
  - University Clinical Center Kragujevac, Kragujevac, Šumadijski Okrug
- Slovakia (2):
  - KM Management, spol. s r.o., Nitra
  - Gastro LM, s.r.o., Prešov
- South Africa (3):
  - CLINRESCO, ARWYP Medical Suites, Johannesburg, Gauteng
  - Dr. J Breedt, Pretoria, Gauteng
  - Dr JP Wright, Claremont, Western Cape
- South Korea (11):
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju, Gang'weondo
  - CHA Bundang Medical Center, CHA University, Seongnam, Gyeonggido
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggido
  - Inje University Haeundae Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Kyungpook National University Chilgok Hospital, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Inje University Seoul Paik Hospital, Seoul
- Spain (9):
  - C.H. Regional Reina Sofia - PPDS, Córdoba, Córdoba
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid, Madrid, Communidad Delaware
  - CHUVI - H.U. Alvaro Cunqueiro, Vigo, Pontevedra
  - Centro Medico Teknon - Grupo Quironsalud, Barcelona
  - Hospital Universitario Juan Ramon Jimenez, Huelva
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
- Mersin University Medical Faculty, Mersin, Turkey (Türkiye)
- Ukraine (13):
  - Regional Municipal Non-profit Enterprise "Chernivtsi Regional Clinical Hospital", Chernivtsi, Chernivtsi Oblast
  - Municipal Nonprofit Enterprise CCH #2 n.a. prof. O.O. Shalimov of Kharkiv City Council, Kharkiv, Kharkivs’ka Oblast’
  - Municipal Non-profit Enterprise of Kyiv Regional Council Kyiv Regional Clinical Hospital, Kyiv, Kyïv
  - LLC Medical Center Family Medicine Clinic, Dnipro
  - Communal Non-Commercial Enterprize of Kharkiv Regional Council Regional Clinical Hospital, Kharkiv
  - Municipal Non-profit Enterprise Kherson City Clinical Hospital named after Ye.Ye. Karabelesh, Kherson
  - Medical Center of LLC Medical Clinic Blagomed, Kyiv
  - Medical Center OK!Clinic+LLC International Institute of Clinical Research, Kyiv
  - Medical Center of LLC Medical Center Dopomoga-Plus, Kyiv
  - Municipal Institution of KRC Kyiv Regional Hospital #2, Kyiv
  - Municipal Nonprofit Enterprise Lviv Clinical Emergency Care Hospital, Lviv
  - Communal Non-Commercial Enterprise Vinnytsia City Clinical Hospital 1, Vinnytsia
  - MNPE City Hospital No. 6 of Zaporizhzhia City Council, Zaporizhzhia
- United Kingdom (4):
  - North Tyneside General Hospital, North Shields, Northumberland
  - Aberdeen Royal Infirmary - PPDS, Aberdeen
  - Royal Gwent Hospital - PPDS, Newport
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Vermeire S, Danese S, Sandborn WJ, Schreiber S, Hanauer S, D'Haens G, Nagy P, Thakur M, Bliss C, Cataldi F, Goetsch M, Gorelick KJ, Reinisch W. Efficacy and Safety of the Anti-mucosal Addressin Cell Adhesion Molecule-1 Antibody Ontamalimab in Patients with Moderate-to-Severe Ulcerative Colitis or Crohn's Disease. J Crohns Colitis. 2024 May 31;18(5):708-719. doi: 10.1093/ecco-jcc/jjad199. PMID 38096402
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fe64db2bf003ab479ae

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 33 sites between 06 February 2019 (first participant first visit) and 13 September 2021 (last participant last visit). 278 sites were initiated in this study, but only 33 sites had enrolled participants.
Pre-assignment Details: A total of 40 participants with moderate to severe Crohn's disease (CD) who completed their participation in an induction study (either SHP647-305 [NCT03559517] or SHP647-306 [NCT03566823]) and fulfilled the efficacy entry criteria of this study, including achieving endoscopic and/or clinical response were enrolled and received study treatment in this study. The study was closed early due to discontinuation of the ontamalimab clinical trial program.
Groups:
- Placebo: Participants received matched placebo of ontamalimab subcutaneous (SC) injection using prefilled syringe on Day 1 Baseline Visit (Week 16 of the SHP647-305 [NCT03559517] or SHP647-306 [NCT03566823]) once every 4 weeks for up to 52 weeks.
- Ontamalimab 25 mg: Participants received 25 mg ontamalimab SC injection, using prefilled syringe on Day 1 Baseline Visit (Week 16 of the SHP647-305 [NCT03559517] or SHP647-306 [NCT03566823]) once every 4 weeks for up to 52 weeks.
- Ontamalimab 75 mg: Participants received 75 mg ontamalimab SC injection, using prefilled syringe on Day 1 Baseline Visit (Week 16 of the SHP647-305 [NCT03559517] or SHP647-306 [NCT03566823]) once every 4 weeks for up to 52 weeks.
Period: Overall Study
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Started | 19 | 10 | 11
Completed | 7 | 4 | 6
Not Completed | 12 | 6 | 5
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 2
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Site terminated by sponsor | 0 | 1 | 0
Not completed — Disease relapse | 7 | 5 | 1
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety set consisted of all participants who have received at least one dose of investigational product (IP) in the SHP647-307 study regardless of treatment received during the induction studies (either SHP647-305 [NCT03559517] or SHP647-306 [NCT03566823]).
Groups:
- Experimental: Ontamalimab 75 mg: Participants received 75 mg ontamalimab SC injection, using prefilled syringe on Day 1 Baseline Visit (Week 16 of the SHP647-305 [NCT03559517] or SHP647-306 [NCT03566823]) once every 4 weeks for up to 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Ontamalimab 25 mg | Experimental: Ontamalimab 75 mg | Total
Number analyzed (Participants) | 19 | 10 | 11 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.7 (14.26) | 38.4 (7.18) | 45.8 (14.85) | 40.1 (13.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 5 | 18
  Male | 12 | 4 | 6 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 3
  Not Hispanic or Latino | 19 | 8 | 10 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 1 | 0 | 0 | 1
  White | 17 | 8 | 10 | 35
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Remission at Week 52
Description: Clinical remission was defined by 2-item PRO sub-scores of average worst daily abdominal pain less than or equal to (<=) 3 (based on 11 point numerical rating scale [NRS] ranging from 0 [no pain] to 10 [worst imaginable pain]); and average daily stool frequency <=2 of type 6/7 (very soft stools/liquid stools) as per the Bristol Stool Form Scale (BSFS) over the 7 most recent days. BSFS ranges from 1 (separate hard lumps, hard to pass), 2 (sausage-shaped, but lumpy), 3 (like a sausage but with cracks on the surface), 4 (like a sausage or snake, smooth and soft), 5 (soft blobs with clear-cut edges), 6 (fluffy pieces with ragged edges, a mushy stool), 7 (watery, no solid pieces, entirely liquid). Participants with missing data at Week 52 or discontinuation before Week 52 were considered failures. Number of participants with clinical remission at Week 52 were reported.
Time Frame: At Week 52
Population: The full analysis set (FAS) consisted of all participants in the randomized set who had received at least 1 dose of investigational product (IP) in the SHP647-307 study regardless of treatment received during the induction studies (either SHP647-305 [NCT03559517] or SHP647-306 [NCT03566823]).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 19 | 10 | 11
Participants | 2 | 3 | 5

2. Primary Outcome: Number of Participants With Enhanced Endoscopic Response at Week 52
Description: Enhanced endoscopic response was defined as a decrease in Simple Endoscopic Score for Crohn's disease (SES-CD) of at least 50 percent (%) from induction study (either SHP647-305 [NCT03559517] or SHP647-306 [NCT03566823] baseline. The SES-CD considers ileum, right colon, transverse colon, left colon, rectum in terms of: size of ulcers, ulcerated surface, affected surface and presence of narrowing. Each graded from 0-3. Scale ranges from 0-56 with a higher score indicating greater severity of disease. Participants with missing data at Week 52 or who discontinued before Week 52 were considered non responders. Number of participants with enhanced endoscopic response at Week 52 were reported.
Time Frame: At Week 52
Population: The FAS consisted of all participants in the randomized set who had received at least 1 dose of IP in the SHP647-307 study regardless of treatment received during the induction studies (either SHP647-305 [NCT03559517] or SHP647-306 [NCT03566823]).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 19 | 10 | 11
Participants | 2 | 4 | 6

3. Secondary Outcome: Number of Participants With Clinical Remission Based on Crohn's Disease Activity Index (CDAI) Score at Week 52
Description: Clinical remission was defined as a CDAI score of <150. CDAI assessed CD based on clinical signs/symptoms such as number of liquid stools, intensity of abdominal pain, general well-being (subjective), and presence of complications, use of antidiarrheal, presence of abdominal mass, physical examination and hematocrit (objective). CDAI score is equal to sum of weighted scores for subjective and objective items which range from 0-149 points: asymptomatic remission, 150-220 points: mild to moderate active CD, 221-450 points: moderate to severe active CD, >451 points: severely active to fulminant disease. Higher score indicating more severity. Participants with missing data at Week 52 or who discontinued before Week 52 were considered failures. Number of participants with clinical remission as measured by CDAI at Week 52 were reported.
Time Frame: At Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 19 | 10 | 11
Participants | 8 | 4 | 7

4. Secondary Outcome: Number of Participants With Glucocorticoid-free Clinical Remission at Week 52
Description: Glucocorticoid-free clinical remission defined as clinical remission by 2-item PRO not requiring any treatment with glucocorticoids for at least 12 weeks prior to Week 52 visit. Clinical remission defined by 2-item PRO sub-scores of average worst daily abdominal pain <=3 (based on 11 point NRS ranging from 0 [no pain] to 10 [worst imaginable pain]); and average daily stool frequency<=2 of type 6/7 (very soft stools/liquid stools) as per the BSFS over the 7 most recent days. BSFS ranges from 1 (separate hard lumps, hard to pass), 2 (sausage-shaped, but lumpy), 3 (like a sausage but with cracks on the surface), 4 (like sausage or snake, smooth and soft), 5 (soft blobs with clear-cut edges), 6 (fluffy pieces with ragged edges, mushy stool), 7 (watery, no solid pieces, entirely liquid). Participants with missing data at Week 52 or who discontinued before Week 52 were non-responders. Number of participants with glucocorticoid-free clinical remission response at Week 52 were reported.
Time Frame: At Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 19 | 10 | 11
Participants | 2 | 1 | 3

5. Secondary Outcome: Number of Participants With Clinical Remission Defined by Crohn's Disease (CD) E-diary Sub-scores- at Week 52
Description: Clinical remission was defined by CD daily e-diary 2-item PRO subscores of average daily abdominal pain <=1 (based on the 4 point scale, with scores ranging from 0 [none] to 3 [severe]) over the 7 most recent days and average daily stool frequency <=3 of type 6/7 (very soft stools/liquid stools) as per the BSFS over the 7 most recent days. BSFS ranges from 1 (separate hard lumps, hard to pass), 2 (sausage-shaped, but lumpy), 3 (like a sausage but with cracks on the surface), 4 (like a sausage or snake, smooth and soft), 5 (soft blobs with clear-cut edges), 6 (fluffy pieces with ragged edges, a mushy stool), 7 (watery, no solid pieces, entirely liquid). Participants with missing data at Week 52 or who discontinued before Week 52 were considered failures. Number of participants with clinical remission based on Crohn's Disease (CD) e-diary Sub-scores for abdominal pain was was reported.
Time Frame: At Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 19 | 10 | 11
Participants | 2 | 3 | 7

6. Secondary Outcome: Number of Participants With Sustained Clinical Remission at Week 52
Description: Sustained clinical remission was defined as clinical remission by 2-item PRO at both Week 52 visit and the maintenance baseline in this Study. Clinical remission was defined by 2-item PRO sub-scores of average worst daily abdominal pain less than or equal to (<=) 3 (based on 11 point NRS ranging from 0 [no pain] to 10 [worst imaginable pain]); and average daily stool frequency <=2 of type 6/7 (very soft stools/liquid stools) as per the BSFS over the 7 most recent days. BSFS ranges from 1 (separate hard lumps, hard to pass), 2 (sausage-shaped, but lumpy), 3 (like a sausage but with cracks on the surface), 4 (like a sausage or snake, smooth and soft), 5 (soft blobs with clear-cut edges), 6 (fluffy pieces with ragged edges, a mushy stool), 7 (watery, no solid pieces, entirely liquid). Number of participants with sustained clinical remission at Week 52 were reported.
Time Frame: At Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 19 | 10 | 11
Participants | 2 | 1 | 2

7. Secondary Outcome: Number of Participants With Sustained Enhanced Endoscopic Response at Week 52
Description: Sustained enhanced endoscopic response was defined as enhanced endoscopic response at both Week 52 visit and the maintenance baseline in this study. Enhanced endoscopic response was defined as a decrease in SES-CD of at least 50 % from induction study (either SHP647-305 [NCT03559517] or SHP647-306 [NCT03566823]) baseline. The SES-CD considers ileum, right colon, transverse colon, left colon, rectum in terms of: size of ulcers, ulcerated surface, affected surface and presence of narrowing. Each graded from 0-3. Scale ranges from 0-56 with a higher score indicating greater severity of disease. Number of participants with sustained enhanced endoscopic response at Week 52 were reported.
Time Frame: At Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 19 | 10 | 11
Participants | 1 | 2 | 3

8. Secondary Outcome: Number of Participants With Clinical Remission Based on 2-item PRO With Enhanced Endoscopic Response at Week 52
Description: Clinical remission was defined by 2-item PRO sub-scores of average worst daily abdominal pain <=3 (based on 11-point NRS) over the 7 most recent days and average daily stool frequency <= 2 of Type 6/7 (very soft stools/liquid stools) as shown in the BSFS over the 7 most recent days. Participants with missing data at Week 52 or who discontinued before Week 52 were considered failures. Enhanced endoscopic response was defined as a decrease in SES-CD of at least 50% from induction study (either SHP647-305 [NCT03559517] or SHP647-306 [NCT03566823]) baseline. Participants with missing data at Week 52 or who discontinued before Week 52 were considered non-responders.
Time Frame: At Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 19 | 10 | 11
Participants | 0 | 3 | 4

9. Secondary Outcome: Number of Participants With Complete Endoscopic Healing at Week 52
Description: Complete endoscopic healing was defined as SES-CD scale score from 0-2. The SES-CD considers ileum, right colon, transverse colon, left colon, rectum in terms of: size of ulcers, ulcerated surface, affected surface and presence of narrowing. Each graded from 0-3. Scale ranges from 0-56 with a higher score indicating greater severity of disease. Participants with missing data at Week 52 or who discontinued before Week 52 were considered failures. Number of participants with complete endoscopic healing at Week 52 were reported.
Time Frame: At Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 19 | 10 | 11
Participants | 0 | 3 | 3

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to 56 weeks
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/10 | 2/11
Other Adverse Events (participants affected / at risk) | 9/19 | 5/10 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | Ontamalimab 25 mg (N=10) | Ontamalimab 75 mg (N=11)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | Ontamalimab 25 mg (N=10) | Ontamalimab 75 mg (N=11)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 3 (4) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroduodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 1 (4)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatic disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Capillary fragility (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The study was closed early as the sponsor discontinued the ontamalimab clinical trial program in CD for reasons unrelated to safety or efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT03627091/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT03627091/SAP_001.pdf